CLINICAL TRIAL: NCT04231019
Title: "Knowledge, Awareness and Perception Regarding Molar-Incisor Hypomineralization Among General Dental Practitioners, Dental Specialists and Dental Students in Egypt"
Brief Title: Knowledge of Egyptian Dental Practitioners Regarding Molar-Incisor Hypomineralization
Acronym: MIH
Status: Completed | Type: Observational
Sponsor: Alaa Mohammed Yehia (Other)
Responsible Party: Sponsor-Investigator, Alaa Mohammed Yehia, Principal Investigator, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: DPH 18-1M
Record Dates: First submitted 2019-12-26; First posted 2020-01-18 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Molar Incisor Hypomineralization; Dental Enamel Hypoplasia
Keywords: Molar incisor hypomineralization; General dental practitioners; Perception; knowledge; Oral health
MeSH Terms: conditions — Molar Hypomineralization; Dental Enamel Hypoplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dental practitioners (general, specialists or students): Two self-administered questionnaires will be used in the study one to general practitioners and specialists and another one with a plain language describing the study will be distributed to the fifth year dental students in Egypt with total 1000 dentist to assess their knowledge, awareness and perception regarding MIH.
  Interventions: Other: self-administered questionnaire

INTERVENTIONS:
Other: self-administered questionnaire — Self-administered questionnaires with plain language statements and brief description of the clinical features and photographs of MIH were used to determine the knowledge, awareness and perception regarding the prevalence, severity, etiology and treatment modalities of molar-incisor hypomineralization (MIH) among Egyptian fifth year dental students, general dental practitioners and dental specialists.
  There were two routes for delivering the questionnaire either as online questionnaire sent to the participants by email or as a hard copy that is hand delivered.

SUMMARY:
Molar incisor hypomineralization (MIH) is one of the developmental enamel defect which is characterized by demarcated, qualitative defects of enamel of systemic origin affecting one to four first permanent molars (FPMs) and frequently associated with incisor involvement. Similar lesions can be seen in second primary molars and their presence has been reported as a predictive factor for developing MIH. Although the exact etiology of MIH is unclear, it is likely to be multi-factorial. Possible etiological factors of MIH are systemic conditions as pneumonia, upper respiratory tract infections, asthma, otitis media, hypoxia, high fever, hypocalcemia and exposure to antibiotics as amoxicillin.

The prevalence of MIH has been reported from several studies to be between 2.8 and 40.2 %, with the mean approximately 15 %. MIH is considered as a common clinical problem by several epidemiological studies from many countries.

Clinical presentation of MIH can include white, creamy and yellow-brown opacities, irregular areas of post eruptive breakdown, which can be mistaken diagnosed as hypoplasia or atypical caries. The condition is usually associated with a high disease burden, leading to pain, infection and tooth loss. Teeth affected by MIH are at high risk of rapid caries development and progression, rapid wear and enamel breakdown. Severely affected enamel disintegrates under masticatory forces resulting in post-eruptive breakdown (PEB), which is also a characteristic feature of MIH-affected teeth. These teeth require treatment, ranging from prevention to restorations and extractions, often under general anesthesia. A multidisciplinary cooperation among clinicians is often required, particularly for extractions of first permanent molars, when orthodontic consequences need to be considered. To evaluate the effect of this condition, questionnaires of dentists and dental professionals have been carried out in various countries, including those in Europe, Australia and New Zealand, Malaysia, Iraq, Iran and Saudi Arabian. These have generally revealed that MIH has been frequently encountered in clinical practice, particularly by dental professionals who treat children and that there is a need for further training for the condition. To date dental clinicians' concerns regarding MIH have not been extensively assessed in Egypt.

DETAILED DESCRIPTION:
In 1970, this condition has been first described as a hypomineralization of the permanent first molars (PFMs) but was consistently referred to it as non-fluoride hypomineralization.

In 2000, there were four presentations that described the same types of developmental defects of dental enamel affecting the first permanent molars (FPM) at the European Academy of Pediatric Dentistry Congress. These reports called the condition hypomineralized first permenet molars FPM, idiopathic enamel hypomineralization in FPM, non-fluoride hypomineralisation in FPM and cheese molars. This was not a new condition. It had been recognized previously but the congress focused on the fact that it has multiple names and that this could conceivably lead to confusion.

In 2001, it has been desirable to use one name that has no reference to any possible etiological factor. So the term "molar-incisor hypomineralization" (MIH) was adopted by Weerheijm to describe these developmental defects and he gave it a definition as "hypomineralization of systemic origin of 1-4 FPM, frequently associated with affected incisors".

In 2003, it was suggested that any examination for MIH should be undertaken on clean wet teeth and optimum at the age of 8-years, as at this age all permanent first molars(PFMs) and most of the incisors will have erupted. The MIH diagnostic criteria are defined using the modified defect of dental enamel (DDE) index, based on criteria by Weerheijm.

Degree of MIH severity Modified DDE index (FDI 1992) Mild degree:- 30% of enamel surface area affected by MIH Moderate degree:- 31 - 49% of enamel surface area affected by MIH Severe degree:- 50% of enamel surface area affected by MIH

Definitions of the criteria used for diagnosing MIH

* Opacity:-A defect involving an alteration in the translucency of the enamel. The defective enamel is of normal thickness at the time of tooth eruption with a smooth surface and white, yellow or brown color. The borders of the lesions are demarcated.
* PEB (post eruptive enamel breakdown):- The defect is indicating deficiency of the surface after eruption of the tooth. This may be caused by such factors as masticatory forces, attrition and trauma (physiological or pathological).
* Atypical Restoration (iatrogenic factor):-Size and shape of restoration do not conform to typical restorative characteristics. In most cases, restorations will be extensive (involving buccal or palatal smooth surface). At the border of the restoration, opacity may be noticed.
* Extraction due to MIH:- Absence of the first permanent molar in a sound dentition is suspected to have been an MIH condition (should take detailed past history, clinical examination of other first permanent molars and incisors).

Many studies have been done to single out a specific etiology for MIH. In 2006, A review by William stated that although an etiology is not known at this time, children who had poor general health in their first three years of life, who were preterm born (low birth weight infants) or were exposed to certain environmental contaminants may be at risk for MIH.

The majority of prevalence and severity studies of MIH to date have taken place in Europe. In 2003, Weerheijm and Mejàre attempted to map its occurrence throughout Europe using a questionnaire sent to members of the European Academy of Pediatric Dentistry.

In 2008, Crombie carried out a questionnaire to assess knowledge of members of the Australian and New Zealand Society of Pediatric Dentistry and found that MIH was widely recognized.

In 2011, a survey mainly about prevalence and etiology of MIH was carried out among teaching staff across all specialties in one dental college in Iraq by Ghanim.

In 2014, two surveys were published investigating the knowledge of Iranian and Malaysian dentists on the etiology, prevalence and management of MIH by Bagheri, Hussein .

In 2014, A study conducted in Jeddah, Saudi Arabia found a prevalence of MIH of 8.6 % by Allazzam and In 2015, another study about the knowledge of Saudi Arabian dental practitioners and students was done by M. J. Silva.

In 2015, A survey was done to estimate the knowledge of pediatric dentists and general dental practitioners in UK.

In 2016, A study on knowledge of Australian and Chilean public oral health care practitioners was done.

The aim of the study is to assess the knowledge of Egyptian dental practitioners regarding the prevalence, etiology, diagnosis and the management of Molar Incisor Hypomineralization (MIH)

ELIGIBILITY:
Inclusion Criteria:

1. Males and females.
2. Dental students should be at the fifth year.
3. All participants should be Egyptians.

Exclusion Criteria:

1. Dentists or dental students who refuse to participate in the study.
2. Any dentist without the Egyptian nationality even if they are studying in Egyptian universities or working in Egypt.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Fifth year dental students, general dental practitioners and dental specialists.
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2018-09-16 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
knowledge of Egyptian dental practitioners regarding molar-incisor hypomineralization | 1 year
  The tool used for measuring the primary outcome is a self-administered questionnaire that was fulfilled by the study participants

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Mo Yehia, Ass. Lec, Principal Investigator — Faculty of Dentistry- Ain Shams University
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Silva MJ, Alhowaish L, Ghanim A, Manton DJ. Knowledge and attitudes regarding molar incisor hypomineralisation amongst Saudi Arabian dental practitioners and dental students. Eur Arch Paediatr Dent. 2016 Aug;17(4):215-22. doi: 10.1007/s40368-016-0230-3. Epub 2016 May 12. PMID 27172776
- [Background] Silva MJ, Scurrah KJ, Craig JM, Manton DJ, Kilpatrick N. Etiology of molar incisor hypomineralization - A systematic review. Community Dent Oral Epidemiol. 2016 Aug;44(4):342-53. doi: 10.1111/cdoe.12229. Epub 2016 Apr 28. PMID 27121068
- [Background] Hussein AS, Ghanim AM, Abu-Hassan MI, Manton DJ. Knowledge, management and perceived barriers to treatment of molar-incisor hypomineralisation in general dental practitioners and dental nurses in Malaysia. Eur Arch Paediatr Dent. 2014 Oct;15(5):301-7. doi: 10.1007/s40368-014-0115-2. Epub 2014 Feb 26. PMID 24569938
- [Background] Ghanim A, Morgan M, Marino R, Manton D, Bailey D. Perception of molar-incisor hypomineralisation (MIH) by Iraqi dental academics. Int J Paediatr Dent. 2011 Jul;21(4):261-70. doi: 10.1111/j.1365-263X.2011.01118.x. Epub 2011 Feb 20. PMID 21332851